CLINICAL TRIAL: NCT04988230
Title: Effects of Time-Restricted Feeding on Nonalcoholic Fatty Liver Disease in Obese Adults: a 12-month Randomized Clinical Trial
Brief Title: Time Restricted Feeding on Nonalcoholic Fatty Liver Disease ( TREATY-FLD )：a 12-month Follow-up Study
Acronym: TREATY-FLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Huijie Zhang, Deputy director of Department of Endocrinology and Metabolism, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFEC-2018-160R
Record Dates: First submitted 2021-07-31; First posted 2021-08-03 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: Nonalcoholic Fatty Liver Disease; Time restricted feeding; Calorie restriction
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Intermittent Fasting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restricted Feeding (Experimental): Participants will receive a diet of 1500-1800kcal/d for men and 1200-1500kcal/d for women during a window of 8 h/d (8 am to 4 pm).
  Interventions: Behavioral: Time restricted feeding
- Continuous Energy Restriction (Active Comparator): Participants will follow receive a diet of 1500-1800kcal/ d for men and 1200-1500kcal/d for women, without restriction on feeding time.
  Interventions: Behavioral: Continuous Energy Restriction

INTERVENTIONS:
Behavioral: Time restricted feeding — Participants will receive a diet of 1500-1800kcal/d for men and 1200-1500kcal/d for women during a window of 8 h/d (8 am to 4 pm).
  Arms: Time Restricted Feeding
Behavioral: Continuous Energy Restriction — Participants will follow receive a diet of 1500-1800kcal/ d for men and 1200-1500kcal/d for women, without restriction on feeding time.
  Arms: Continuous Energy Restriction

SUMMARY:
Time restricted feeding (TRF) is a novel type of intermittent calorie restriction diet that involves eating a daily period of 8 hours or less. This is a 6-month follow-up study of TREATY-FLD trial to evaluate the effect of time restricted feeding (TRF) on hepatic fat contents and cardiometabolic risk factors in obese adults over 6 months compared to continuous energy restriction (CER).

ELIGIBILITY:
Inclusion Criteria:

1. Man or women aged≥18 years;
2. Subjects with NAFLD determined by MRI (intrahepatic triglyceride content ≥5%);
3. Body mass index (BMI)of 28.0 to 45.0 kg/m2;

Exclusion Criteria:

1. History of alcoholic liver disease, chronic viral hepatitis, drug-induced hepatitis, autoimmune hepatitis, cirrhosis, and liver cancer;
2. History of HIV, or active pulmonary tuberculosis;
3. Diagnosis of type 1 and type 2 diabetes;
4. History of malignant tumors;
5. Serious liver dysfunction or chronic kidney disease (AST or ALT > 3 times the upper limit of normal, or eGFR<30 ml/min/1.73 m2);
6. Significant alcohol consumption in the past six months (Consumed more than 20 g/day for women or 30 g/day for men);
7. History of serious cardiovascular or cerebrovascular disease (angina, myocardial infarction or stroke) in the past 6 months;
8. History of severe gastrointestinal diseases or gastrointestinal surgery in the past 12 months;
9. History of Cushing's syndrome, hypothyroidism, acromegaly, hypothalamic obesity;
10. Being a smoker or having been a smoker in the 3 months prior to their screening visit;
11. Taking medications affecting weight or energy intake/energy expenditure in the last 6 months, including weight loss medications, antipsychotic drugs or other medications as determined by the study physician;
12. Currently participating in weight loss programs or weight change in the past 3 months (> 5% current body weight) ;
13. Women who are pregnant or plan to become pregnant;
14. Patients who cannot be followed for 24 months (due to a health situation or migration);
15. Patients who are unwilling or unable to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Change in intrahepatic fat content | Baseline,month 6, month 12.
  Intrahepatic fat content will be assessed by MR mDixon-Quant

SECONDARY OUTCOMES:
Change in liver fiber | Baseline,month 6, month 12.
  Liver fiber will be assessed by liver Fibrotouch
Change in visceral fat | Baseline,month 6, month 12.
  Visceral fat will be assessed by abdominal CT scan
Change in body fat | Baseline,month 6, month 12.
  Body fat will be assessed by whole-body dual x-ray system
Change in waist circumference | Baseline,month 6, month 12.
Change in body weight | Baseline,month 6, month 12.
Change in HbA1c level | Baseline,month 6, month 12.
Change in Systolic blood pressure | Baseline,month 6, month 12.
Change in LDL-c level | Baseline,month 6, month 12.
Change in serum ALT level | Baseline,month 6, month 12.
Change in insulin sensitivity | Baseline,month 6, month 12.
  Insulin sensitivity will be assessed by HOMA-IR

CONTACTS AND LOCATIONS:
Overall Officials: Huijie Zhang, MD,PhD, Study Chair — Department of Endocrinology and Metabolism, Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wei X, Lin B, Huang Y, Yang S, Huang C, Shi L, Liu D, Zhang P, Lin J, Xu B, Guo D, Li C, He H, Liu S, Xue Y, Xu Y, Zhang H. Effects of Time-Restricted Eating on Nonalcoholic Fatty Liver Disease: The TREATY-FLD Randomized Clinical Trial. JAMA Netw Open. 2023 Mar 1;6(3):e233513. doi: 10.1001/jamanetworkopen.2023.3513. PMID 36930148